CLINICAL TRIAL: NCT00100815
Title: Multicenter, Open Label, Phase II Clinical Study of Gemcitabine, Capecitabine and Avastin in Pancreatic Cancer
Brief Title: Gemcitabine, Capecitabine, and Bevacizumab in Treating Patients With Metastatic or Unresectable Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000409556; RPCI-I-19903; GENENTECH-RPCI-I-19903
Record Dates: First submitted 2005-01-06; First posted 2005-01-07 (Estimated); Results first posted 2015-12-24 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-11

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; recurrent pancreatic cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Bevacizumab; Capecitabine; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: bevacizumab — 30-90 minutes on day 1, every 21 days up to 12 months.
Drug: capecitabine — twice daily on days 1-14. Courses repeat every 21 days for up to 12 months in the absence of disease progression or unacceptable toxicity.
Drug: gemcitabine hydrochloride — IV over 30 minutes on days 1 and 8. Courses repeat every 21 days for up to 12 months in the absence of disease progression or unacceptable toxicity.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Bevacizumab may stop the growth of tumor cells by stopping blood flow to the tumor. Giving gemcitabine and capecitabine together with bevacizumab may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving gemcitabine and capecitabine together with bevacizumab works in treating patients with metastatic or unresectable pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine progression-free survival of patients with metastatic or unresectable adenocarcinoma of the pancreas treated with gemcitabine, capecitabine, and bevacizumab.

Secondary

* Determine clinical response in patients treated with this regimen.
* Determine toxicity of this regimen in these patients.
* Determine quality of life of patients treated with this regimen.

OUTLINE: This is an open-label, multicenter study.

Patients receive bevacizumab IV over 30-90 minutes on day 1, oral capecitabine twice daily on days 1-14, and gemcitabine IV over 30 minutes on days 1 and 8. Courses repeat every 21 days for up to 12 months in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline then weekly for 3 weeks.

Patients are followed every 2-4 months for 1 year and then every 6 months for at least 5 years.

PROJECTED ACCRUAL: A total of 35 patients will be accrued for this study within 8.8-17.5 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the pancreas meeting 1 of the following criteria:

  * Newly diagnosed or previously treated metastatic disease
  * Unresectable disease
* No CNS or brain metastases

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* ECOG 0-1

Life expectancy

* More than 3 months

Hematopoietic

* Absolute neutrophil count > 1,500/mm^3
* WBC > 3,000/mm^3
* Platelet count > 100,000/mm^3
* Hemoglobin ≥ 9 g/dL (transfusion or epoetin alfa allowed)
* No evidence of bleeding diathesis or coagulopathy

Hepatic

* Bilirubin < 2 mg/dL
* AST or ALT < 2.5 times upper limit of normal (ULN) (5 times ULN if liver metastases are present)
* INR < 1.5 (except for patients receiving full-dose warfarin)

Renal

* Creatinine < 1.5 mg/dL
* No proteinuria OR
* Urine protein < 500 mg by 24-hour urine collection
* No clinically significant impairment of renal function

Cardiovascular

* No uncontrolled hypertension (blood pressure > 160/110 mm Hg on medication)
* No New York Heart Association class II-IV congestive heart failure
* No unstable symptomatic arrhythmia requiring medication

  * Chronic atrial arrhythmia (i.e., atrial fibrillation or paroxysmal supraventricular tachycardia) allowed
* No clinically significant grade II-IV peripheral vascular disease
* No arterial thromboembolic event within the past 6 months, including any of the following:

  * Transient ischemic attack
  * Cerebrovascular accident
  * Unstable angina
  * Myocardial infarction

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other serious systemic disease
* No significant traumatic injury within the past 28 days
* No serious non-healing wound, ulcer, or bone fracture
* No history of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* More than 28 days since prior major surgery or open biopsy
* More than 7 days since prior fine needle aspirations or core biopsies
* No concurrent major surgery

Other

* More than 4 weeks since prior and no concurrent participation in any other experimental drug study
* More than 12 months since prior adjuvant therapy
* No prior systemic therapy for metastatic disease

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2004-08; Primary Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renuka Iyer, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (2):
- United States (2):
  - Roswell Park Cancer Institute, Buffalo, New York
  - Case Comprehensive Cancer Center, Cleveland, Ohio

REFERENCES:
- [Result] Javle M, Yu J, Garrett C, Pande A, Kuvshinoff B, Litwin A, Phelan J 3rd, Gibbs J, Iyer R. Bevacizumab combined with gemcitabine and capecitabine for advanced pancreatic cancer: a phase II study. Br J Cancer. 2009 Jun 16;100(12):1842-5. doi: 10.1038/sj.bjc.6605099. Epub 2009 Jun 2. PMID 19491904

RESULTS

PARTICIPANT FLOW:
Groups:
- GEMCITABINE, CAPECITABINE and AVASTIN: Avastin 15 mg/ kg q 3 weeks, starting day 1; capecitabine 650 mg/m2 bid x 14 days starting day 1, gemcitabine 1000 mg/m2 days 1 and 8, cycles to be repeated q 21 days.
Period: Overall Study
Arm/Group | GEMCITABINE, CAPECITABINE and AVASTIN
Started | 50
Completed | 1
Not Completed | 49
Not completed — Progression | 24
Not completed — Adverse Event | 18
Not completed — Death | 4
Not completed — Other | 3

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Arm/Group | GEMCITABINE, CAPECITABINE and AVASTIN
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.18 (11.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 28

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progressive Disease is defined using the international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee [JNCI 92(3):205-216, 2000], as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of one or more new lesions, or appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: every 2-4 months for 1 year and then every 6 months for 5 years
Population: All treated and eligible patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | GEMCITABINE, CAPECITABINE and AVASTIN
Number analyzed (Participants) | 50
months | 5.7 [4.2 to 7.2]

2. Secondary Outcome: Percentage of Participants With Grades 3-5 Treatment Related Toxicities
Description: Grade 3, 4 or 5 toxicity rate
Time Frame: Subjects were evaluated for adverse events at each study visit for the duration of their participation in the study, up to 5 years
Population: All treated and eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GEMCITABINE, CAPECITABINE and AVASTIN
Number analyzed (Participants) | 50
percentage of participants | 70 [55.4 to 82.1]

3. Secondary Outcome: Percentage of Participants With Improved Quality of Life
Description: Quality of Life was assessed using EORTC QLQ-PAN26. All measures range in score from 1 to 4 as lower scores indicate better outcomes. The improved Quality of Life is defined as a greater than 5% decrease in 2 consecutive scores compared with the baseline score.
Time Frame: assessed at baseline then weekly for 3 weeks
Population: All treated and eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GEMCITABINE, CAPECITABINE and AVASTIN
Number analyzed (Participants) | 50
percentage of participants | 56.0 [41.3 to 70.0]

4. Secondary Outcome: Clinical Response
Description: Response was evaluated using the international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee [JNCI 92(3):205-216, 2000]. Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), At least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter; Overall Response (OR) = CR + PR.
Time Frame: Pre-treatment and every 6 weeks from treatment.
Population: All treated and eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GEMCITABINE, CAPECITABINE and AVASTIN
Number analyzed (Participants) | 50
percentage of participants | 22.0 [11.5 to 35.9]

5. Secondary Outcome: Overall Survival
Time Frame: every 2-4 months for 1 year and then every 6 months for 5 years
Population: All treated and eligible patients
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | GEMCITABINE, CAPECITABINE and AVASTIN
Number analyzed (Participants) | 50
months | 9.8 [8.3 to 12.6]

ADVERSE EVENTS:
Arm/Group | GEMCITABINE, CAPECITABINE and AVASTIN
Serious Adverse Events (participants affected / at risk) | 27/50
Other Adverse Events (participants affected / at risk) | 47/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GEMCITABINE, CAPECITABINE and AVASTIN (N=50)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3)
Myocardial infarction (Cardiac disorders) | 1 (1)
Blindness (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (5)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (5)
Asthenia (General disorders) | 1 (1)
Death (General disorders) | 5 (5)
Device occlusion (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1)
Pain (General disorders) | 3 (3)
Pyrexia (General disorders) | 5 (6)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Febrile infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (2)
Haemoglobin (Investigations) | 1 (1)
Neutrophil count (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 4 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Balance disorder (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Female genital tract fistula (Reproductive system and breast disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 2 (2)
Haemorrhage (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GEMCITABINE, CAPECITABINE and AVASTIN (N=50)
Anaemia (Blood and lymphatic system disorders) | 18 (29)
Leukopenia (Blood and lymphatic system disorders) | 6 (9)
Lymphopenia (Blood and lymphatic system disorders) | 3 (4)
Neutropenia (Blood and lymphatic system disorders) | 16 (31)
Spleen disorder (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (16)
Arrhythmia (Cardiac disorders) | 1 (1)
Cardiomegaly (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Eye swelling (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 13 (14)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Chapped lips (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 13 (16)
Diarrhoea (Gastrointestinal disorders) | 17 (24)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 3 (3)
Faecaloma (Gastrointestinal disorders) | 1 (1)
Faeces discoloured (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 3 (3)
Gastric varices (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 1 (1)
Gingival polyp (Gastrointestinal disorders) | 1 (1)
Glossodynia (Gastrointestinal disorders) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 21 (28)
Oesophagitis (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 5 (6)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 7 (13)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 11 (12)
Asthenia (General disorders) | 4 (5)
Chest pain (General disorders) | 3 (3)
Chills (General disorders) | 7 (7)
Device occlusion (General disorders) | 4 (4)
Fatigue (General disorders) | 30 (44)
Influenza like illness (General disorders) | 2 (2)
Local swelling (General disorders) | 1 (1)
Mucosal inflammation (General disorders) | 3 (3)
Oedema (General disorders) | 11 (15)
Oedema peripheral (General disorders) | 4 (5)
Pain (General disorders) | 12 (14)
Pyrexia (General disorders) | 9 (14)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (3)
Cellulitis (Infections and infestations) | 1 (1)
Cystitis (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 2 (2)
Influenza (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (2)
Wound complication (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 11 (18)
Antineutrophil cytoplasmic antibody (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 13 (25)
Blood albumin (Investigations) | 15 (18)
Blood albumin decreased (Investigations) | 4 (4)
Blood alkaline phosphatase (Investigations) | 16 (31)
Blood alkaline phosphatase increased (Investigations) | 3 (3)
Blood amylase increased (Investigations) | 1 (1)
Blood bicarbonate (Investigations) | 6 (6)
Blood bilirubin (Investigations) | 10 (18)
Blood bilirubin increased (Investigations) | 1 (2)
Blood calcium (Investigations) | 8 (10)
Blood chloride (Investigations) | 5 (6)
Blood creatinine (Investigations) | 7 (7)
Blood creatinine decreased (Investigations) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Blood glucose (Investigations) | 6 (18)
Blood lactate dehydrogenase (Investigations) | 4 (5)
Blood lactate dehydrogenase increased (Investigations) | 1 (1)
Blood potassium (Investigations) | 12 (19)
Blood potassium increased (Investigations) | 1 (1)
Blood pressure (Investigations) | 6 (8)
Blood sodium (Investigations) | 7 (8)
Blood urea (Investigations) | 6 (6)
Blood uric acid decreased (Investigations) | 4 (5)
Blood uric acid increased (Investigations) | 4 (4)
Carbon dioxide abnormal (Investigations) | 1 (1)
Creatinine renal clearance (Investigations) | 1 (2)
Haematocrit (Investigations) | 6 (7)
Haemoglobin (Investigations) | 20 (30)
Haemoglobin decreased (Investigations) | 2 (2)
International normalised ratio (Investigations) | 4 (5)
International normalised ratio increased (Investigations) | 1 (1)
Lipase (Investigations) | 1 (1)
Liver function test (Investigations) | 1 (1)
Lymphocyte count (Investigations) | 1 (2)
Lymphocyte count abnormal (Investigations) | 1 (1)
Neutrophil count (Investigations) | 17 (31)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count (Investigations) | 13 (20)
Platelet count decreased (Investigations) | 5 (6)
Platelet count increased (Investigations) | 2 (3)
Protein total (Investigations) | 4 (5)
Protein total decreased (Investigations) | 3 (3)
Protein urine (Investigations) | 1 (1)
Prothrombin time prolonged (Investigations) | 1 (1)
Red blood cell count (Investigations) | 11 (14)
Urine output increased (Investigations) | 1 (1)
Weight (Investigations) | 1 (1)
Weight decreased (Investigations) | 13 (17)
White blood cell count (Investigations) | 16 (22)
White blood cell count abnormal (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 5 (6)
White blood cell count increased (Investigations) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 16 (18)
Dehydration (Metabolism and nutrition disorders) | 7 (9)
Hyperalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 21 (30)
Hyperkalaemia (Metabolism and nutrition disorders) | 5 (6)
Hypernatraemia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 (16)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Ageusia (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 9 (9)
Dysarthria (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 4 (5)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Depressed mood (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 3 (3)
Dysphoria (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 4 (5)
Restlessness (Psychiatric disorders) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 2 (2)
Proteinuria (Renal and urinary disorders) | 2 (3)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (11)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 8 (14)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 6 (6)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Yellow skin (Skin and subcutaneous tissue disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2)
Hot flush (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 16 (27)
Hypotension (Vascular disorders) | 5 (6)
Orthostatic hypotension (Vascular disorders) | 3 (3)
Phlebitis (Vascular disorders) | 1 (1)
Subclavian vein thrombosis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes